CLINICAL TRIAL: NCT02615613
Title: Effect of Food Acceptability on Appetite Hormones' Response in Normal Weight Male Subjects
Brief Title: The Effect of Food Hedonics on Appetite Hormones Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Ammar Olabi, Associate Professor, American University of Beirut Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NUT.AO.11
Record Dates: First submitted 2015-11-25; First posted 2015-11-26 (Estimated); Last update posted 2015-11-30 (Estimated); Status verified 2015-11

CONDITIONS: Eating Behavior
Keywords: Hedonics, Ghrelin, Hunger
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High acceptability meal (Experimental): A custard recipe was used as the high acceptability meal
  Interventions: Other: High acceptability meal
- Low acceptability meal (Experimental): The regular custard recipe was reformulated to yield a low acceptability version
  Interventions: Other: Low Acceptability Meal

INTERVENTIONS:
Other: Low Acceptability Meal
  Arms: Low acceptability meal
Other: High acceptability meal
  Arms: High acceptability meal

SUMMARY:
30-40 healthy male subjects with a BMI between 18.5 and 24.9 kg/m2 will be tested for food preferences using a questionnaire with 141 different foods. Accordingly, a high acceptability/palatability food will be selected (average score of ≥ 7 on the 9-point hedonic scale). Two versions of the selected high palatability food will be devised by modifying it to yield the original high and the modified low acceptability versions. The two versions will differ only in palatability and will be equicaloric. Subjects who agree on the acceptability of the two versions of the food (11 subjects) will consume, at fasting, the two versions of the food in a cross over design over two sessions. Each session will include an acceptability test, using the 9-point hedonic scale, on three instances: after sampling a spoonful, eating the whole portion and after 240 min. The quantity consumed on each session will constitute 30% of the subject's resting energy expenditure. Moreover, fasting and postprandial hunger ratings and blood samples will be collected at time 0 and after 15, 30, 60, 120, 180 and 240 min of the food/meal's ingestion. The visual analogue scale will be used for huger ratings.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Male
* Age: 18-50 years
* Body Mass Index (BMI): 18.5-24.9 kg/m2
* Stable body weight for at least three months before the study with absence of any form of dieting, food restriction or other abnormal eating behaviors (to minimize effect of weight change on ghrelin status)

Exclusion Criteria:

* Smoking
* Substance abuse such as alcohol or drugs
* Medical or psychological illness
* Use of medications
* Previous gastrointestinal surgery
* History of weight fluctuation (weight loss of greater than 5% within the past 3 months)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Food acceptability score | Two weeks
Ghrelin level | Two weeks

SECONDARY OUTCOMES:
Glucose level | Two weeks
Appetite score on the visual analogue scale | Two weeks
Insulin level | 2 weeks